CLINICAL TRIAL: NCT03376347
Title: HYPE Trial. Intraoperative Implementation of the Hypotension Probability Indicator (HPI) Algorithm: a Pilot Randomized Controlled Clinical Trial
Brief Title: Intraoperative Implementation of the Hypotension Probability Indicator
Acronym: HYPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, D.P.Veelo, Principal Investigator, Medical Doctor, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL 6211501817
Record Dates: First submitted 2017-12-03; First posted 2017-12-18 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Intraoperative Hypotension
Keywords: intraoperative; hypotension; Hypotension Probability Index; HPI
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional arm (No Intervention): Institutional Standard of Care with intention to keep MAP> 65 mmHg. The FlotracIQ will be connected, but fully covered.
- Treatment arm (Active Comparator): FlotracIQ with HPI algorithm.
  Interventions: Device: FlotracIQ with HPI algorithm

INTERVENTIONS:
Device: FlotracIQ with HPI algorithm — FlotracIQ with hypotension probability indicator (HPI) algorithm connected to arterial line. The treating anesthetist is provided with guidance by means of a flowchart suggesting when to treat and what. Timing of treatment and choice of treatment is then left to the discretion of the attending physician.
  Arms: Treatment arm

SUMMARY:
Reducing intraoperative hypotension using FlotracIQ with HPI software.

DETAILED DESCRIPTION:
Intraoperative hypotension occurs often. Even short durations of hypotension are suggested to be associated with increased risk for renal insufficiency and myocardial ischemia. Currently treatment of these hypotensive episodes is not proactive. Edwards Lifesciences has developed an algorithm using continuous invasively-measured arterial waveforms to predict hypotension with high accuracy minutes before blood pressure actually decreases. Hypothesis: the use of this algorithm will alter treatment of hypotension and reduces the incidence of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Planned for elective non-cardiac non-day surgery with an expected duration of more than 2 hours
* Planned to receive general anaesthesia
* Planned to receive an arterial line during surgery
* Aim for MAP of 65 mmHg during surgery
* Being able to give written informed consent prior to surgery

Exclusion Criteria:

* Aim for MAP other than 65 mmHg at discretion treating physician
* Significant hypotension before surgery defined as a MAP <65
* Right- or left sided cardiac failure (e.g. LVEF<35%)
* Known cardiac shunts (significant)
* Known aortic stenosis (severe)
* Severe cardiac arrhythmias including atrial fibrillation
* Requiring dialysis
* Liver surgery
* Vascular surgery with clamping of the aorta
* Perioperative Goal Directed Therapy (PGDT) protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
TWA hypotension (measured with FlotracIQ) | intraoperative, starting 15 minutes after induction
  Time weighted average spent in hypotension, defined as MAP <65mmHg for ≥1min

SECONDARY OUTCOMES:
Incidence of hypotension (measured with FlotracIQ) | intraoperative, starting 15 minutes after induction
  Incidence of hypotension, defined as MAP <65mmHg for ≥1min
Time spent in hypotension (measured with FlotracIQ) | intraoperative, starting 15 minutes after induction
  Time spent in hypotension, in minutes, defined as MAP <65mmHg for ≥1min
TWA hypertension (measured with FlotracIQ) | intraoperative, starting 15 minutes after induction
  Time weighted average spent in hypertension, defined as MAP >100 mmHg for ≥1min
Percentage of time in hypertension (measured with FlotracIQ) | intraoperative, starting 15 minutes after induction
  Percentage of time in hypertension, defined as MAP >100 mmHg for ≥1min
Incidence of hypertension (measured with FlotracIQ) | intraoperative, starting 15 minutes after induction
  Incidence of hypertension, defined as MAP >100 mmHg for ≥1min.
Treatment choice (CRF, EPD) | intraoperative, starting 15 minutes after induction
  Medication used to prevent/treat hypotension. A study member is present at the OR to make notes
Treatment dose (CRF, EPD) | intraoperative, starting 15 minutes after induction
  Dose of medication used to prevent/treat hypotension. A study member is present at the OR to make notes
Time to treatment (CRF) | intraoperative, starting 15 minutes after induction
  time to treatment of hypotension, defined as MAP <65mmHg for ≥1min. A study member is present at the OR to make notes
Diagnostic guidance protocol deviations (CRF) | intraoperative, starting 15 minutes after induction
  Diagnostic guidance protocol deviations, a study member is present at the OR to make notes of any protocol deviations.

CONTACTS AND LOCATIONS:
Overall Officials: M.W. Hollmann, MD, PhD, Principal Investigator — Academic Medical Center (AMC), Amsterdam
Locations (1):
- Academic Medical Center Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827
- [Derived] Wijnberge M, Schenk J, Terwindt LE, Mulder MP, Hollmann MW, Vlaar AP, Veelo DP, Geerts BF. The use of a machine-learning algorithm that predicts hypotension during surgery in combination with personalized treatment guidance: study protocol for a randomized clinical trial. Trials. 2019 Oct 11;20(1):582. doi: 10.1186/s13063-019-3637-4. PMID 31601239